CLINICAL TRIAL: NCT02047331
Title: Multimodal Periarticular Injection Versus Fascia Iliaca Compartment Block for Total Knee Arthroplasty
Brief Title: Periarticular Injection Versus Fascia Iliaca Block for Total Knee Arthroplasty
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, CAGLA BALI,MD, MD,Anesthesiology and Reanimation, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA12/269
Record Dates: First submitted 2014-01-23; First posted 2014-01-28 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Total Knee Arthroplasty
Keywords: periarticular drug injection; fascia iliaca block; knee arthroplasty

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group PI (Active Comparator): group PI were performed periarticular drug injection during surgery.
  Interventions: Procedure: periarticular injection
- group FI (Active Comparator): group FI were performed fascia iliaca block before surgery
  Interventions: Procedure: fascia iliaca block

INTERVENTIONS:
Procedure: periarticular injection — patients were performed bupivacaine solution to the periarticular soft tissues during surgery by the surgeon.
  Arms: group PI
Procedure: fascia iliaca block — patients were performed fascia iliaca block with bupivacaine solution before surgery.
  Arms: group FI

SUMMARY:
In this study, the aim is to compare the efficacy of Periarticular multimodal drug injection(group PI) and Fascia Iliaca Compartment Block ( group FI)for total knee arthroplasty.

DETAILED DESCRIPTION:
Total knee arthroplasty is very painful surgical intervention.Patients were assigned to 2 groups to receive either periarticular multimodal drug injection or fascia iliaca compartment block for postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing knee arthroplasty
* > 18 years of age

Exclusion Criteria:

* obesity
* heart failure
* kidney failure
* liver failure

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Postoperative pain scores of periarticular injection and fascia block for total knee arthroplasty | postoperative 24 hours
  Patients were assigned in two groups to perform either periarticular injection (group PI) and fascia block ( group FB). They were accessed by visual analog scale. The aim was to compare the efficacy and side effects of periarticular injection and fascia block.

CONTACTS AND LOCATIONS:
Overall Officials: Anis Aribogan, Prof.,MD, Study Director — Baskent University School of Medicine
Locations (1):
- Baskent University School of Medicine Adana Teaching and reserach Hospital, Adana, Turkey (Türkiye)